CLINICAL TRIAL: NCT05123495
Title: Safe Introduction of a New Surgical Device With the Device Briefing Tool and Surgical Safety Checklist in Singapore
Brief Title: Device Briefing Tool and Surgical Safety Checklist Implementation
Status: Completed | Type: Observational
Sponsor: James Etheridge (Other)
Collaborators: Singapore General Hospital (Other)
Responsible Party: Sponsor-Investigator, James Etheridge, Safe Surgery Research Fellow, Ariadne Labs
Organization: Ariadne Labs (Other)
Other Study IDs: IRB19-0389
Record Dates: First submitted 2021-10-18; First posted 2021-11-17 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Clinical Skills
Keywords: Non-technical skills

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Device Briefing Tool Implementation: Surgical departments which receive training on use of the Device Briefing Tool
  Interventions: Behavioral: Device Briefing Tool; Behavioral: Surgical Safety Checklist
- Comparator: Surgical departments that do not receive training on use of the Device Briefing Tool
  Interventions: Behavioral: Surgical Safety Checklist

INTERVENTIONS:
Behavioral: Device Briefing Tool — A 4-item supplement to the WHO Surgical Safety Checklist designed to improve teamwork and communication around new/complex surgical devices
  Groups: Device Briefing Tool Implementation
Behavioral: Surgical Safety Checklist — Reimplementation of the WHO Surgical Safety Checklist to improve adherence and utility of the checklist

SUMMARY:
The investigators aim to implement a quality improvement initiative using the device briefing tool (DBT) and the Safe Surgery Checklist (SSC) and to evaluate its effect on patient safety measures and on safety culture with the introduction of a new surgical device in Singapore hospitals. Within eligible hospitals, J&J and Ariadne Labs staff will train local implementation teams to, in turn, train operating room teams to use the DBT and SSC. Project-specific outcomes will be measured by neutral observers and via survey data. Throughout the quality improvement initiative, hospitals will receive ongoing training and coaching on their interventions and feedback on their outcomes.

DETAILED DESCRIPTION:
Design of Quality Improvement Initiative Using a prospective observational implementation design, surgical teams will be assigned to 1 of 2 groups. Group I will receive the complete intervention, which includes implementation of the DBT from the start, and then the DBT and SSC package.

Group II does not receive the DBT alone; these teams continue with their usual care, and then receive the DBT and SSC package.

Device-related interruptions, non-technical skills of surgical teams, and Culture of Safety Survey will be measured pre- and post-implementation of the SSC and DBT interventions, with specific timing depended on group allocation. OR teams at each hospital will be observed longitudinally to assess the effects of the DBT and SSC interventions.

Target Population for the Quality Improvement Initiative Participants will be members of the OR team at each participating hospital. These members include practicing surgeons, anesthesiologists, OR nurses, and OR staff. Hospitals will be participating institutions of SingHealth and NUHS hospital clusters. J&J device sales representatives ("reps") will serve as key trainers during the multidisciplinary trainings to use the DBT during an operation. A separate implementation team will be trained by Ariadne Labs to execute the SSC at each eligible hospital. Hospital leadership will be key stakeholders to engage at each hospital in order to implement the DBT, team training, and SSC program.

Interventions Device Briefing Tool: a 4-item mini-checklist focused on raising OR team awareness to the nuances of a new surgical device.

Trained J&J sales reps will be responsible for training OR teams to use the DBT with the new surgical device. Ariadne Labs will provide initial training to the J&J reps and be available for ongoing training support.

Safe Surgery Checklist: Developed with the World Health Organization, the SSC is a 19-item checklist consisting of verbal confirmation by surgical teams of the completion of the basic steps for ensuring the safe delivery of anesthesia, prophylaxis against infection, effective teamwork, among other essential practices in surgery. As described elsewhere in greater detail, it is used at 3 critical junctures of care: before anesthesia is administered, immediately before incision is made, and before the patient is taken out of the operating room. A successful implementation of the SSC is a labor-intensive iterative process that includes 4 phases: prepare, own, expand, and improve.

Ariadne Labs will provide the specialists needed to implement the SSC and to support local hospitals' implementation teams. Please refer to the SSC Implementation Guide for process details in the Supplemental Materials.

Outcomes to Study Device-related interruptions: Any interruption in the surgical team's workflow as the result of the use of the study device.

Non-technical skills: Evaluation of OR team performance for non-technical skills (situation awareness, decision-making, cooperation and teamwork, and leadership), using the NOTECHS assessment, a validated rating system for intraoperative OR team behavior.

Perception of safety, i.e. "safety culture": The perception of safety among members of the OR team will be measured using the Culture of Safety Survey.

Site readiness assessment: We will evaluate the readiness capacity of institutions to implement the DBT/SSC intervention using the Readiness Assessment Tool.

Goal: Determine if the pre-intervention Readiness Assessment Tool is predictive (R2 > 0.7) of implementation success as gauged by the post-intervention Implementation Survey.

Feasibility of scale: The scale of this project will be measured by the number of personnel trained, the number of hospitals at which the DBT, team training, and SSC intervention is implemented, and adherence rates to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Surgical teams in SingHealth hospitals

Exclusion Criteria:

* Refusal by any team member to participate

Note - there are NO specific age criteria, since the unit of analysis is the surgical team rather than the patient. It is highly unlikely that any surgical team member would be less than 18 years of age or greater than 89 years of age, but there are no explicit age-based exclusions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All surgical teams operating in participating SingHealth hospitals will be eligible. Surgical teams include surgeons, anesthetists, nurses, and (in some cases) ancillary providers. The patient is not included as a member of the surgical team. Patients are not being evaluated as part of this study.
Sampling Method: Non-Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Oxford NOTECHS scale | Change in NOTECHS scores will be assessed from baseline to immediately after DBT implementation and 2-months after SSC implementation
  Measure of non-technical skills of surgical teams assessed by neutral observers. Scored 12-48 with higher scores indicating better non-technical skills.

SECONDARY OUTCOMES:
Device-related interruptions (DRIs) | Change in DRIs will be assessed from baseline to immediately after DBT implementation and 2-months after SSC implementation
  The number of times surgical teams must cease activity due to a problem with a surgical device
Culture of safety | Change in safety culture from baseline will be assessed 2-months post-SSC
  Safety culture, as measured by division-wide Hospital Survey on Patient Safety Culture (HSOPS) survey. HSOPS is scored from 0 to 100% with higher scores indicating better safety culture.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim Havens, MD, Principal Investigator — Ariadne Labs
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No